CLINICAL TRIAL: NCT05889611
Title: Iterative Endotracheal Tube Cuff Pressure Monitoring
Acronym: SIPBIE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8904
Record Dates: First submitted 2023-05-22; First posted 2023-06-05 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Spine Disease
Keywords: Spine Disease; Spine surgery; Intubation Cuff Pressure; Endotracheal Intubation; Upper airways
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Studies in the medical literature underline the importance of monitoring the pressure of the balloon and the relationship with the incidence cited on the pain and discomfort related to the gesture of the upper airways. There are no formal recommendations in the literature, the French Society of Anesthesia and Resuscitation (SFAR) recommends monitoring the pressure intraoperatively except after intubation. It would be interesting to see and thus make an inventory of the practices, to reiterate the importance of monitoring throughout the gesture and at the change of position to avoid either micro-inhalation linked to under pressure of the balloon or overpressure which causes a potential risk of tracheal injury.

ELIGIBILITY:
Inclusion criteria:

* Elderly patient ≥ 18 years old
* Patient who has a scheduled spine intervention in the prone position from January 1, 2023 to April 30, 2023
* Intubated patient with endotracheal tube under mechanical ventilation
* Sedation and curarization
* ASA 1, 2 and 3
* Duration of surgery > 1 hour
* Subject not objecting to the reuse of their data for the purposes of this research.

Exclusion criteria:

* Subject who expressed their opposition to participating in the study
* ASA 4, difficult intubation and emergency
* Lung pathologies (asthma, COPD, tracheomalacia)
* Severe heart failure
* Septic, cardiogenic or volume shock
* Morbid obesity (BMI >40)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient who has a scheduled spine intervention in the prone position from January 1, 2023 to April 30, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-03-22 (Estimated); Study Completion 2024-03-22 (Estimated)

PRIMARY OUTCOMES:
Balloon pressure | Throughout the surgical procedure
  Monitoring of balloon pressure following prone position during spine surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas PARTOUCHE, MD, Study Director — University Hospitals of Strasbourg
Locations (1):
- Service d'Anesthésiologie - Réanimation Chirurgicale - CHU de Strasbourg - France, Strasbourg, France